CLINICAL TRIAL: NCT03351296
Title: Randomized Phase 2 Trial Of Two Chemotherapy Regimens Plus Or Minus Bevacizumab In Patients With Well Differentiated Pancreatic Neuroendocrine Tumors
Brief Title: Two Chemotherapy Regimens Plus or Minus Bevacizumab
Acronym: BETTER2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-000741-46; 2017/2523 (Other: CSET number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Streptozocin; Capecitabine; Temozolomide; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Comparative phase II trial with two randomizations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LV5FU2 + streptozotocin (Experimental)
  Interventions: Drug: LV5FU2; Drug: Streptozocin
- Capecitabine + temozolomide (Experimental)
  Interventions: Drug: Capecitabine; Drug: Temozolomide
- LV5FU2 + streptozotocin + Bevacizumab (Experimental)
  Interventions: Drug: LV5FU2; Drug: Streptozocin; Drug: Bevacizumab
- Capecitabine + temozolomide + Bevacizumab (Experimental)
  Interventions: Drug: Capecitabine; Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Drug: LV5FU2 — LV5FU2 (Folinic Acid D, L 400 mg/m² day 1, 5FU 400 mg/m² IV bolus, 5FU 2400 mg/m² 48 hours continuous infusion)
  Arms: LV5FU2 + streptozotocin; LV5FU2 + streptozotocin + Bevacizumab
Drug: Streptozocin — streptozotocin 800 mg/m² day 1 every 14 days
  Arms: LV5FU2 + streptozotocin; LV5FU2 + streptozotocin + Bevacizumab
Drug: Capecitabine — Capecitabine 750 mg/m² twice daily, days 1-14
  Arms: Capecitabine + temozolomide; Capecitabine + temozolomide + Bevacizumab
Drug: Temozolomide — temozolomide 200 mg/m² once daily, days 10-14, every 28 days
  Arms: Capecitabine + temozolomide; Capecitabine + temozolomide + Bevacizumab
Drug: Bevacizumab — bevacizumab 5 mg/kg every 14 days
  Arms: Capecitabine + temozolomide + Bevacizumab; LV5FU2 + streptozotocin + Bevacizumab

SUMMARY:
Compare the effect of capecitabine (cape) + temozolomide (temo) and of 5FU + streptozotocin (strepto) given with a new schedule (LV5FU2 + strepto), two of the most used chemotherapy regimens in the treatment of well differentiated pancreatic neuroendocrine tumors alone or in combination with bevacizumab (beva) on progression-free survival (PFS) and compare the chemotherapy regimens alone or with beva (two by two design) on the same criteria.

ELIGIBILITY:
1. Well differentiated pancreatic neuroendocrine tumor grade 1 (NET G1), grade 2 (NET G2) or grade 3 (NET G3)*

   *Grade 3 tumor must be confirmed by a pathologist of the TENpath network.
2. Indication for chemotherapy for locally advanced or metastatic disease with proven progression (at least 20% increase of tumor size on a maximum of 12 months period of follow-up) or other indication of chemotherapy following the National Thesaurus of GI Cancerology (Appendix 6) (liver involvement > 50%, symptoms related to the tumour or its metastases, Ki67>10%)
3. Patient with at least one measurable target tumor by RECIST 1.1 and that has never been irradiated
4. Patient with a life expectancy greater than 3 months
5. Men or women with performance status (ECOG) ≤ 2 (Appendix 3)
6. Age ≥ 18 years
7. Adequate hematological function: neutrophil count (ANC) ≥ 1.5x109/L, platelets greater than 75x109/L, hemoglobin greater than 10g/dl (blood transfusions are accepted to reach this level).
8. Adequate liver function: serum bilirubin lower than 3 x upper limit of normal (ULN); aminotransferases and alkaline phosphatase levels lower than 2.5 ULN (lower than 5 ULN if liver metastases), TP greater than 50 %
9. Proteinuria lower than 1g/24h, blood creatinine less than 120 μmol/L and creatinin clearance ≥ 60 ml/min as calculated by Cockroft-Gault formula Note: a negative dipstick urine analysis is sufficient.
10. Absence of active bleeding, coagulopathy or pathologic condition that would confer a high risk of bleeding
11. Prior treatment with somatostatin analogues, everolimus or sunitinib is allowed
12. Negative serum pregnancy test ≤ 72 hours before randomization (for women of childbearing potential only). Sexually active women of childbearing potential must agree to use a highly effective method of contraception or to abstain from sexual activity during the study and for at least 6 months after the last study treatment administration. Sexually active males patients must agree to use condom during the study and for at least 6 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception.
13. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
14. Patient affiliated to a social security regimen or beneficiary of such regimen

Non inclusion criteria :

1. Disease accessible to resection or percutaneous method of destruction
2. Any known allergy or contraindication to the treatments used in the trial
3. Patients with a complete DPD deficiency; defined as an uracil concentration ≥150ng/ml Note: patients with a suspicion of partial DPD deficiency, defined as a uracil concentration ≥ 16 ng/ml and < 150 ng/ml, will receive an adapted 1st cycle dose, according to a clinic-biological discussion. The dose can be then readapted for the second cycle according to the tolerability of the treatment during the 1st cycle.
4. Patient previously treated with chemotherapy for the neuroendocrine tumour
5. Patient have received any other antitumor therapy: chemotherapy, immunotherapy
6. Other serious diseases such as respiratory failure or congestive heart failure, angina pectoris not medically controlled; history of myocardial infarction within 6 months prior to study entry, uncontrolled hypertension and arrhythmias, concomitant severe infection or uncontrolled diabetes mellitus
7. Subjects with a history of chronic or acute hepatitis C or B infection.
8. Surgery during the 5 weeks preceding the randomization
9. History of cancer (except basal cell skin or carcinoma in situ carcinoma of the cervix) within 5 years prior to entry into the trial. But patients with cancers that have been treated more than 5 years ago and are considered as cured are eligible.
10. Neurological or psychiatric pathology that may interfere with adherence to treatment
11. Patients have received yellow fever vaccine within 30 days prior to the first dose of trial treatment.
12. Patient with pernicious anaemia and other megaloblastic anaemias secondary to the lack of Vitamin B12
13. Hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies
14. Hypersensitivity to study drugs or any of its excipients
15. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
16. Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate | Until disease progression or unacceptable toxicity (median 24 months)

SECONDARY OUTCOMES:
Toxicity (NCI-CTCAE 4.0) | Until disease progression or unacceptable toxicity

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - CHU de Caen, Caen, Calvados
  - CHU de Dijon, Dijon, Côte d'Or
  - Hôpital Haut-Lévêque, Pessac, Gironde
  - IUCT - Hôpital Rangueil, Toulouse, Haute-Garonne
  - Hôpital Beaujon, Clichy, Hauts-de-Seine
  - ICM Val d'Aurelle, Montpellier, Hérault
  - Hôpital Trousseau CHU Tours, Chambray-lès-Tours, Indre-et-Loire
  - Institut de Cancérologie de l'Ouest site René Gauducheau, Saint-Herblain, Loire-Atlantique
  - CHR d'Orléans, Orléans, Loiret
  - CHU Angers, Angers, Maine-et-Loire
  - Hôpital Haut-Lévêque, Reims, Marne
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hôpital Edouard Herriot, Lyon, Rhône
  - Gustave Roussy, Villejuif, Val De Marne
  - Hôpital Croix St Simon, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Eugène Marquis, Rennes, Île-et-Vilaine

IPD SHARING:
Plan to Share IPD: Undecided